CLINICAL TRIAL: NCT00387088
Title: Efficacy {FEV1, COPD Exacerbations & HRQoL} & Safety of 5mcg Tiotropium Respimat in COPD
Brief Title: Tiotropium / Respimat One Year Study in COPD.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 205.372; 2006-001009-27
Record Dates: First submitted 2006-10-11; First posted 2006-10-12 (Estimated); Results first posted 2010-01-22 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2013-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

ARMS (2):
- Tiotropium (Other): Tiotropium 5µg via Respimat® inhaler (2 inhalations of 2.5µg per day) + usual maintenance treatment (only anticholinergic bronchodilators were excluded)
  Interventions: Drug: Tiotropium
- Placebo (Other): Placebo via Respimat® inhaler (2 inhalations per day) + usual maintenance treatment (only anticholinergic bronchodilators were excluded)
  Interventions: Device: Respimat

INTERVENTIONS:
Device: Respimat
  Arms: Placebo
Drug: Tiotropium
  Arms: Tiotropium

SUMMARY:
The objective of the study is to evaluate the long-term (one year) efficacy and safety of tiotropium delivered by the Respimat inhaler in patients with COPD. Specifically, the study will examine the effect of treatment on COPD exacerbations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. At least 40 years old
3. Smoker or ex-smoker
4. Smoking history > 10 pack-years
5. Forced Expiratory Volume in 1 Second (FEV1) < 60% predicted

Exclusion Criteria:

1. Recent history of myocardial infarction, life-threatening cardiac arrhythmia or hospitalisation for cardiac failure
2. History of asthma or allergic conditions.
3. Malignancy requiring treatment within past 5 years
4. Life-threatening pulmonary obstruction, cystic fibrosis or clinically evident bronchiectasis
5. Known active tuberculosis
6. Known hypersensitivity to anticholinergic drugs.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3991 (Actual)
Dates: Start 2006-09; Primary Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (334):
- United States (57):
  - 205.372.01012 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 205.372.01020 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 205.372.01062 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 205.372.01048 Boehringer Ingelheim Investigational Site, Berkeley, California
  - 205.372.01037 Boehringer Ingelheim Investigational Site, Huntington Park, California
  - 205.372.01058 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 205.372.01059 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 205.372.01007 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 205.372.01034 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 205.372.01028 Boehringer Ingelheim Investigational Site, Rancho Mirage, California
  - 205.372.01011 Boehringer Ingelheim Investigational Site, San Diego, California
  - 205.372.01066 Boehringer Ingelheim Investigational Site, Boulder, Colorado
  - 205.372.01008 Boehringer Ingelheim Investigational Site, Norwalk, Connecticut
  - 205.372.01004 Boehringer Ingelheim Investigational Site, Brandon, Florida
  - 205.372.01060 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 205.372.01069 Boehringer Ingelheim Investigational Site, Miami Beach, Florida
  - 205.372.01023 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 205.372.01053 Boehringer Ingelheim Investigational Site, Winter Park, Florida
  - 205.372.01045 Boehringer Ingelheim Investigational Site, Calhoun, Georgia
  - 205.372.01043 Boehringer Ingelheim Investigational Site, Normal, Illinois
  - 205.372.01061 Boehringer Ingelheim Investigational Site, Dubuque, Iowa
  - 205.372.01035 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 205.372.01049 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 205.372.01015 Boehringer Ingelheim Investigational Site, Biddeford, Maine
  - 205.372.01067 Boehringer Ingelheim Investigational Site, Columbia, Maryland
  - 205.372.01006 Boehringer Ingelheim Investigational Site, Rockville, Maryland
  - 205.372.01013 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 205.372.01003 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 205.372.01021 Boehringer Ingelheim Investigational Site, Chesterfield, Missouri
  - 205.372.01014 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 205.372.01036 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 205.372.01046 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 205.372.01024 Boehringer Ingelheim Investigational Site, Mineola, New York
  - 205.372.01029 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 205.372.01030 Boehringer Ingelheim Investigational Site, Syracuse, New York
  - 205.372.01026 Boehringer Ingelheim Investigational Site, Chapel Hill, North Carolina
  - 205.372.01019 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 205.372.01027 Boehringer Ingelheim Investigational Site, Elizabeth City, North Carolina
  - 205.372.01038 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 205.372.01031 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 205.372.01017 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 205.372.01041 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 205.372.01044 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 205.372.01001 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 205.372.01063 Boehringer Ingelheim Investigational Site, Eugene, Oregon
  - 205.372.01068 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 205.372.01056 Boehringer Ingelheim Investigational Site, Swathmore, Pennsylvania
  - 205.372.01039 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 205.372.01050 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 205.372.01005 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 205.372.01018 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 205.372.01040 Boehringer Ingelheim Investigational Site, New Braunfels, Texas
  - 205.372.01052 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 205.372.01022 Boehringer Ingelheim Investigational Site, Danville, Virginia
  - 205.372.01065 Boehringer Ingelheim Investigational Site, Lynchburg, Virginia
  - 205.372.01055 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 205.372.01064 Boehringer Ingelheim Investigational Site, Tacoma, Washington
- Australia (10):
  - 205.372.61002 Woolcock Institute of Medical Research, Glebe, New South Wales
  - 205.372.61009 Thoracic & General Physician, Cairns, Queensland
  - 205.372.61005 Redcliffe Hospital, Redcliffe, Queensland
  - 205.372.61006 The Investigator Clinic, Port Lincoln, South Australia
  - 205.372.61007 The Burnside War Memorial Hospital, Toorak Gardens, South Australia
  - 205.372.61004 Boehringer Ingelheim Investigational Site, Woodville, South Australia
  - 205.372.61010 Ecru, Box Hill, Victoria
  - 205.372.61008 Geelong Clinical Research Centre, Geelong, Victoria
  - 205.372.61001 Emeritus Research, Malvern, Victoria
  - 205.372.61003 Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Brazil (6):
  - 205.372.55012 Universidade Federal de Santa Catarina, Florianópolis
  - 205.372.55009 Hospital das Clínicas de Goiânia, Goiânia
  - 205.372.55005 Hospital Geral Otávio de Freitas, Recife
  - 205.372.55001 INCOR e Hospital das Clínicas da Universidade de São Paulo, São Paulo - SP
  - 205.372.55010 Unidade de Coracao e Pulmao do Dto. de Medicina, São Paulo - SP
  - 205.372.55011 CEDOES - Diagnóstico e Pesquisa, Vitória
- Canada (19):
  - 205.372.11007 Heritage Medical Research Building, Calgary, Alberta
  - 205.372.11013 Calgary West Medical Centre, Calgary, Alberta
  - 205.372.11011 Hermitage Medicentre, Edmonton, Alberta
  - 205.372.11017 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 205.372.11020 Wetaskiwin Lung Laboratory, Wetaskiwin, Alberta
  - 205.372.11010 Dr. Kay Ho, Chilliwack, British Columbia
  - 205.372.11018 Pacific Lung Health Centre, Vancouver, British Columbia
  - 205.372.11005 Professional Corp. Respirology, Saint John, New Brunswick
  - 205.372.11009 White Hills Medical Clinic, St. John's, Newfoundland and Labrador
  - 205.372.11012 West Lincoln Memorial Hospital, Grimsby, Ontario
  - 205.372.11014 Dr. Robert Luton, London, Ontario
  - 205.372.11001 Niagara Clinical Research, Niagara Falls, Ontario
  - 205.372.11019 Allergy and Asthma Research Centre, Ottawa, Ontario
  - 205.372.11003 London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - 205.372.11016 London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - 205.372.11002 Centenary Respiratory Research Associates, Scarborough Village, Ontario
  - 205.372.11006 Clinique de médecine familiale de La Malbaie, La Malbaie, Quebec
  - 205.372.11004 Mount Royal Family Physicians, Saskatoon, Saskatchewan
  - 205.372.11015 Dr. Arun Nayar, Saskatoon, Saskatchewan
- China (12):
  - 205.372.86002 Boehringer Ingelheim Investigational Site, Beijing
  - 205.372.86003 Boehringer Ingelheim Investigational Site, Beijing
  - 205.372.86004 Boehringer Ingelheim Investigational Site, Beijing
  - 205.372.86009 Boehringer Ingelheim Investigational Site, Chengdu, Sichuan Province
  - 205.372.86008 Boehringer Ingelheim Investigational Site, Chongqing
  - 205.372.86001 Boehringer Ingelheim Investigational Site, Guangzhou
  - 205.372.86010 Boehringer Ingelheim Investigational Site, Shanghai
  - 205.372.86011 Boehringer Ingelheim Investigational Site, Shanghai
  - 205.372.86012 Boehringer Ingelheim Investigational Site, Shanghai
  - 205.372.86005 Boehringer Ingelheim Investigational Site, Shenyang
  - 205.372.86006 Boehringer Ingelheim Investigational Site, Shenyang
  - 205.372.86007 Boehringer Ingelheim Investigational Site, Wuhan
- Denmark (6):
  - 205.372.45004 Boehringer Ingelheim Investigational Site, Aarhus C
  - 205.372.45005 Boehringer Ingelheim Investigational Site, Horsens
  - 205.372.45002 Boehringer Ingelheim Investigational Site, Hvidovre
  - 205.372.45001 Boehringer Ingelheim Investigational Site, København NV
  - 205.372.45003 Boehringer Ingelheim Investigational Site, Odense C
  - 205.372.45006 Boehringer Ingelheim Investigational Site, Silkeborg
- Finland (4):
  - 205.372.35804 Boehringer Ingelheim Investigational Site, Helsinki
  - 205.372.35802 Boehringer Ingelheim Investigational Site, Jyväskylä
  - 205.372.35803 Boehringer Ingelheim Investigational Site, Lahti
  - 205.372.35801 Boehringer Ingelheim Investigational Site, Tampere
- France (28):
  - 205.372.3318A Clinique du Parc, Castelnau-le-Lez
  - 205.372.3318B Clinique du Parc, Castelnau-le-Lez
  - 205.372.3304A Cabinet Médical, Chamalières
  - 205.372.3301A Hôpital Gabriel Montpied, Clermont-Ferrand
  - 205.372.3310A Centre Hospitalier, Denain
  - 205.372.3314A Cabinet Médical, Grasse
  - 205.372.3306A Hôpital Ambroise Paré, Marseille
  - 205.372.3303A Hôpital Notre Dame de Bon Secours, Metz
  - 205.372.3303B Hôpital Notre Dame de Bon Secours, Metz
  - 205.372.3312A Cabinet Médical, Montigny-lès-Metz
  - 205.372.3312B Cabinet Médical, Montigny-lès-Metz
  - 205.372.3302A Centre Médical Erdre Saint Augustin, Nantes
  - 205.372.3305A Cabinet Médical, Nice
  - 205.372.3305B Cabinet Médical, Nice
  - 205.372.3315A Hôpital Caremeau, Nîmes
  - 205.372.3315B Hôpital Caremeau, Nîmes
  - 205.372.3317A Cabinet de Pneumologie, Nîmes
  - 205.372.3320A Polyclinique Les Fleurs, Ollioules
  - 205.372.3320B Polyclinique Les Fleurs, Ollioules
  - 205.372.3316A Clinique les Bleuets, Reims
  - 205.372.3316B Clinique les Bleuets, Reims
  - 205.372.3321A Centre Hospitalier, Saint-Gaudens
  - 205.372.3321C Centre Hospitalier, Saint-Gaudens
  - 205.372.3319A Institut Arnault Tzanck, Saint-Laurent-du-Var
  - 205.372.3325A Cabinet Médical, Six Four Les Plages
  - 205.372.3324A Cabinet Médical, Toulon
  - 205.372.3309A Cabinet médical, Toulouse
  - 205.372.3309B Cabinet médical, Toulouse
- Germany (16):
  - 205.372.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 205.372.49004 Boehringer Ingelheim Investigational Site, Berlin
  - 205.372.49013 Boehringer Ingelheim Investigational Site, Berlin
  - 205.372.49007 Boehringer Ingelheim Investigational Site, Bonn
  - 205.372.49008 Boehringer Ingelheim Investigational Site, Bruchsal
  - 205.372.49011 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 205.372.49012 Boehringer Ingelheim Investigational Site, Gelnhausen
  - 205.372.49006 Boehringer Ingelheim Investigational Site, Gütersloh
  - 205.372.49014 Boehringer Ingelheim Investigational Site, Hanover
  - 205.372.49005 Boehringer Ingelheim Investigational Site, Kassel
  - 205.372.49009 Boehringer Ingelheim Investigational Site, Minden
  - 205.372.49010 Boehringer Ingelheim Investigational Site, München
  - 205.372.49016 Boehringer Ingelheim Investigational Site, Weinheim
  - 205.372.49015 Boehringer Ingelheim Investigational Site, Weyhe
  - 205.372.49001 Boehringer Ingelheim Investigational Site, Wiesloch
  - 205.372.49003 Boehringer Ingelheim Investigational Site, Witten
- Greece (15):
  - 205.372.30001 Boehringer Ingelheim Investigational Site, Athens
  - 205.372.30002 Boehringer Ingelheim Investigational Site, Athens
  - 205.372.30003 Boehringer Ingelheim Investigational Site, Athens
  - 205.372.30013 Boehringer Ingelheim Investigational Site, Athens
  - 205.372.30015 Boehringer Ingelheim Investigational Site, Athens
  - 205.372.30011 Boehringer Ingelheim Investigational Site, Corinth
  - 205.372.30009 Boehringer Ingelheim Investigational Site, Heraklion-Crete
  - 205.372.30007 Boehringer Ingelheim Investigational Site, Kalamaria
  - 205.372.30005 Boehringer Ingelheim Investigational Site, Kavala
  - 205.372.30004 Boehringer Ingelheim Investigational Site, Komotini
  - 205.372.30019 Boehringer Ingelheim Investigational Site, Nafplion
  - 205.372.30008 Boehringer Ingelheim Investigational Site, Serres
  - 205.372.30014 Boehringer Ingelheim Investigational Site, Thebes
  - 205.372.30006 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 205.372.30017 Boehringer Ingelheim Investigational Site, Thessaloniki
- Hong Kong (2):
  - 205.372.85203 Boehringer Ingelheim Investigational Site, Hong Kong
  - 205.372.85201 Boehringer Ingelheim Investigational Site, Kowloon
- Hungary (6):
  - 205.372.36001 Boehringer Ingelheim Investigational Site, Budapest
  - 205.372.36002 Boehringer Ingelheim Investigational Site, Debrecen
  - 205.372.36004 Boehringer Ingelheim Investigational Site, Deszk
  - 205.372.36005 Boehringer Ingelheim Investigational Site, Érd
  - 205.372.36006 Boehringer Ingelheim Investigational Site, Mosonmagyaróvár
  - 205.372.36007 Boehringer Ingelheim Investigational Site, Sopron
- India (17):
  - 205.372.91005 Boehringer Ingelheim Investigational Site, Andhra Pradesh
  - 205.372.91016 Boehringer Ingelheim Investigational Site, Andhra Pradesh
  - 205.372.91003 Boehringer Ingelheim Investigational Site, Bangalore
  - 205.372.91006 Boehringer Ingelheim Investigational Site, Bangalore
  - 205.372.91017 Boehringer Ingelheim Investigational Site, Calicut,Kerala
  - 205.372.91007 Boehringer Ingelheim Investigational Site, Chennai
  - 205.372.91010 Boehringer Ingelheim Investigational Site, Chennai
  - 205.372.91002 Boehringer Ingelheim Investigational Site, Coimbatore
  - 205.372.91009 Boehringer Ingelheim Investigational Site, Gujarat
  - 205.372.91011 Boehringer Ingelheim Investigational Site, indore,MP
  - 205.372.91012 Boehringer Ingelheim Investigational Site, Maharashtra
  - 205.372.91004 Boehringer Ingelheim Investigational Site, Mumbai
  - 205.372.91008 Boehringer Ingelheim Investigational Site, Mumbai
  - 205.372.91015 Boehringer Ingelheim Investigational Site, New Delhi
  - 205.372.91014 Boehringer Ingelheim Investigational Site, Punjab
  - 205.372.91013 Boehringer Ingelheim Investigational Site, Tamil Nadu
  - 205.372.91001 Boehringer Ingelheim Investigational Site, Uttar Pradesh
- 205.372.35303 Boehringer Ingelheim Investigational Site, Mullingar, Ireland
- Italy (12):
  - 205.372.39007 Boehringer Ingelheim Investigational Site, Bussolengo (vr)
  - 205.372.39012 Boehringer Ingelheim Investigational Site, Ferrara
  - 205.372.39003 Boehringer Ingelheim Investigational Site, Genova
  - 205.372.39004 Boehringer Ingelheim Investigational Site, Genova
  - 205.372.39005 Boehringer Ingelheim Investigational Site, Milan
  - 205.372.39008 Boehringer Ingelheim Investigational Site, Modena
  - 205.372.39009 Boehringer Ingelheim Investigational Site, Orbassano (to)
  - 205.372.39001 Boehringer Ingelheim Investigational Site, Pisa
  - 205.372.39010 Boehringer Ingelheim Investigational Site, Pordenone
  - 205.372.39002 Boehringer Ingelheim Investigational Site, Prato (fi)
  - 205.372.39011 Boehringer Ingelheim Investigational Site, Roma
  - 205.372.39006 Boehringer Ingelheim Investigational Site, Trieste
- Lithuania (3):
  - 205.372.37001 Boehringer Ingelheim Investigational Site, Kaunas
  - 205.372.37003 Boehringer Ingelheim Investigational Site, Kaunas
  - 205.372.37002 Boehringer Ingelheim Investigational Site, Vilnius
- Malaysia (7):
  - 205.372.60003 Boehringer Ingelheim Investigational Site, George Town
  - 205.372.60007 Boehringer Ingelheim Investigational Site, Johor Bahru
  - 205.372.60004 Boehringer Ingelheim Investigational Site, Kelantan Darul Naim
  - 205.372.60005 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 205.372.60006 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 205.372.60001 Boehringer Ingelheim Investigational Site, Kuala Selangor
  - 205.372.60002 Boehringer Ingelheim Investigational Site, Kuching, Sarawak
- Mexico (14):
  - 205.372.52018 Hospital Universitario de Chihuahua, Chihuahua City
  - 205.372.52017 Instituto Nacional de Enfermedades Respiratorias (INER), Col. Seccion XVI
  - 205.372.52013 Sanatorio Henri Dunant, Cuernavaca, Mor. México
  - 205.372.52005 Hospital Civil Nuevo de Guadalajara, Guadalajara
  - 205.372.52009 Hospital Civil Antiguo, Guadalajara Jal.
  - 205.372.52001 Hospital General del Estado de Sonora, Hermosillo, Sonora
  - 205.372.52014 Hospital Angeles de las Lomas, Huixquilucan Edo.Mex.
  - 205.372.52004 Clínica de Mérida, Merida Yuc.
  - 205.372.52016 Hospital General de Mexicali, Mexicali Baja California Norte
  - 205.372.52010 Hospital General Agustin O´Haran, Mérida Yucatán
  - 205.372.52002 Unidad de Investigación clínica en Medicina, Monterrey, Nuevo León
  - 205.372.52006 Hospital Universitario, Monterrey, Nuevo León
  - 205.372.52012 Hospital de Nuestra Señora de la Salud, San Luis Potosí City
  - 205.372.52003 Hospital "Angel Leaño", Zapopan, Jal.
- Netherlands (11):
  - 205.372.31009 Boehringer Ingelheim Investigational Site, Amsterdam
  - 205.372.31006 Boehringer Ingelheim Investigational Site, Drachten
  - 205.372.31001 Boehringer Ingelheim Investigational Site, Groningen
  - 205.372.31011 Boehringer Ingelheim Investigational Site, Hoofddorp
  - 205.372.31007 Boehringer Ingelheim Investigational Site, Leeuwarden
  - 205.372.31004 Boehringer Ingelheim Investigational Site, Roosendaal
  - 205.372.31003 Boehringer Ingelheim Investigational Site, Sneek
  - 205.372.31012 Boehringer Ingelheim Investigational Site, Utrecht
  - 205.372.31002 Boehringer Ingelheim Investigational Site, Voorburg
  - 205.372.31008 Boehringer Ingelheim Investigational Site, Weerselo
  - 205.372.31005 Boehringer Ingelheim Investigational Site, Winschoten
- Norway (3):
  - 205.372.47002 Boehringer Ingelheim Investigational Site, Ålesund
  - 205.372.47001 Boehringer Ingelheim Investigational Site, Sandvika
  - 205.372.47003 Boehringer Ingelheim Investigational Site, Trondheim
- Portugal (5):
  - 205.372.35102 Hospital Fernando Fonseca, Amadora
  - 205.372.35101 Hospital Pulido Valente, Lisbon
  - 205.372.35104 Hospital de Santa Marta, Lisbon
  - 205.372.35103 Hospital de São João, Porto
  - 205.372.35105 Centro Hospitalar do Alto Minho, Estrada de Santa Luzia, Viana do Castelo
- Singapore (3):
  - 205.372.65001 Boehringer Ingelheim Investigational Site, Singapore
  - 205.372.65003 Boehringer Ingelheim Investigational Site, Singapore
  - 205.372.65005 Boehringer Ingelheim Investigational Site, Singapore
- Slovakia (2):
  - 205.372.42102 Boehringer Ingelheim Investigational Site, Bratislava
  - 205.372.42103 Boehringer Ingelheim Investigational Site, Nové Zámky
- South Africa (8):
  - 205.372.27002 Boehringer Ingelheim Investigational Site, Bellville
  - 205.372.27001 Boehringer Ingelheim Investigational Site, Cape Town
  - 205.372.27004 Boehringer Ingelheim Investigational Site, Cape Town
  - 205.372.27008 Boehringer Ingelheim Investigational Site, Cape Town
  - 205.372.27006 Boehringer Ingelheim Investigational Site, Centurion
  - 205.372.27003 Boehringer Ingelheim Investigational Site, Durban
  - 205.372.27005 Boehringer Ingelheim Investigational Site, Pretoria
  - 205.372.27007 Boehringer Ingelheim Investigational Site, Somerset West
- South Korea (10):
  - 205.372.82010 Boehringer Ingelheim Investigational Site, Anyang
  - 205.372.82005 Boehringer Ingelheim Investigational Site, Daegu
  - 205.372.82009 Boehringer Ingelheim Investigational Site, Daejoen
  - 205.372.82003 Boehringer Ingelheim Investigational Site, Incheon
  - 205.372.82008 Boehringer Ingelheim Investigational Site, Jeonbuk
  - 205.372.82007 Boehringer Ingelheim Investigational Site, Kwangju
  - 205.372.82002 Boehringer Ingelheim Investigational Site, Pusan
  - 205.372.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 205.372.82004 Boehringer Ingelheim Investigational Site, Seoul
  - 205.372.82006 Boehringer Ingelheim Investigational Site, Seoul
- Spain (5):
  - 205.372.34005 Hospital San Pedro de Alcántara, Cáceres
  - 205.372.34004 Hospital Gregorio Marañón, Madrid
  - 205.372.34006 Hospital 12 de octubre, Madrid
  - 205.372.34001 Hospital Mutua Terrassa, Terrassa (Barcelona)
  - 205.372.34002 Hospital Universitario Dr. Peset, Valencia
- Sweden (5):
  - 205.372.46001 Björknäs Vårdcentral, Boden
  - 205.372.46004 Näsets läkargrupp, Höllviken
  - 205.372.46005 Lungmedicinska kliniken, Linköping
  - 205.372.46006 Lungmedicinska Kliniken, Stockholm
  - 205.372.46002 Alnö Vårdcentral, Sundsvall
- Switzerland (3):
  - 205.372.41002 Boehringer Ingelheim Investigational Site, Lugano
  - 205.372.41003 Boehringer Ingelheim Investigational Site, Montana
  - 205.372.41001 Boehringer Ingelheim Investigational Site, Zurich
- Taiwan (9):
  - 205.372.88607 Kaohsiung Medical University Hospital, Kaohsiung City
  - 205.372.88606 National Cheng Kung University Hospital, Tainan
  - 205.372.88601 National Taiwan University Hospital, Taipei
  - 205.372.88602 Taipei Veterans General Hospital, Taipei
  - 205.372.88603 Mackay Memorial Hospital, Taipei
  - 205.372.88604 Tri-Service General Hospital, Taipei
  - 205.372.88608 Boehringer Ingelheim Investigational Site, Taipei
  - 205.372.88609 Boehringer Ingelheim Investigational Site, Taipei
  - 205.372.88605 Chang Gung Memorial Hosp-Linkou, Taoyuan District
- Turkey (Türkiye) (10):
  - 205.372.90006 Gazi Universitesi Tip Fakultesi Gogus Hastaliklari A.B.D., Ankara
  - 205.372.90007 Atatürk Gög. Hastaliklari ve Cerrahisi Egitim Hastanesi, Ankara
  - 205.372.90003 Uludag Universitesi Tip Fakultesi Gogus Hastaliklari, Bursa
  - 205.372.90009 Trakya Universitesi Tip Fakultesi Gogus Hastaliklari A.B.D., Edirne
  - 205.372.90004 Dr. Lütfi Kirdar Egitim ve Arastirma Hastanesi, Istanbul
  - 205.372.90005 Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - 205.372.90001 Izmir Tepecik Gogus Hastaliklari ve Gogus Cerrahisi Hast., Izmir
  - 205.372.90008 Erciyes Universitesi Tip Fakultesi, Kayseri
  - 205.372.90010 Selcuk Universitesi Tip Fakultesi, Konya
  - 205.372.90002 19 Mayis Universitesi Tip Fakultesi Gogus Hastaliklari A.B.D, Samsun
- United Kingdom (25):
  - 205.372.44027 Boehringer Ingelheim Investigational Site, Aston Clinton, Aylesbury
  - 205.372.44022 Boehringer Ingelheim Investigational Site, Carmarthen
  - 205.372.44002 Boehringer Ingelheim Investigational Site, Chertsey
  - 205.372.44023 Boehringer Ingelheim Investigational Site, Chesterfield
  - 205.372.44014 Boehringer Ingelheim Investigational Site, Darlington
  - 205.372.44009 Boehringer Ingelheim Investigational Site, East Horsley
  - 205.372.44011 Boehringer Ingelheim Investigational Site, Fowey
  - 205.372.44003 Boehringer Ingelheim Investigational Site, Frome
  - 205.372.44026 Boehringer Ingelheim Investigational Site, Greenisland
  - 205.372.44013 Boehringer Ingelheim Investigational Site, Heywood
  - 205.372.44016 Boehringer Ingelheim Investigational Site, Isleworth
  - 205.372.44020 Boehringer Ingelheim Investigational Site, Kirkby in Ashfield
  - 205.372.44024 Boehringer Ingelheim Investigational Site, Mortimer
  - 205.372.44001 Boehringer Ingelheim Investigational Site, Nottingham
  - 205.372.44018 Boehringer Ingelheim Investigational Site, Penzance
  - 205.372.44021 Boehringer Ingelheim Investigational Site, Plymouth
  - 205.372.44005 Boehringer Ingelheim Investigational Site, Saint Just, Penzance
  - 205.372.44007 Boehringer Ingelheim Investigational Site, Sheffield
  - 205.372.44010 Boehringer Ingelheim Investigational Site, Sneinton, Nottingham
  - 205.372.44015 Boehringer Ingelheim Investigational Site, St Austell
  - 205.372.44006 Boehringer Ingelheim Investigational Site, Sunderland
  - 205.372.44008 Boehringer Ingelheim Investigational Site, Wellingborough
  - 205.372.44012 Boehringer Ingelheim Investigational Site, Westbury on Trym
  - 205.372.44028 Boehringer Ingelheim Investigational Site, Windsor
  - 205.372.44019 Boehringer Ingelheim Investigational Site, Woking

REFERENCES:
- [Derived] Singh D, Wedzicha JA, Siddiqui S, de la Hoz A, Xue W, Magnussen H, Miravitlles M, Chalmers JD, Calverley PMA. Blood eosinophils as a biomarker of future COPD exacerbation risk: pooled data from 11 clinical trials. Respir Res. 2020 Sep 17;21(1):240. doi: 10.1186/s12931-020-01482-1. PMID 32943047
- [Derived] Bateman ED, Tashkin D, Siafakas N, Dahl R, Towse L, Massey D, Pavia D, Zhong NS. A one-year trial of tiotropium Respimat plus usual therapy in COPD patients. Respir Med. 2010 Oct;104(10):1460-72. doi: 10.1016/j.rmed.2010.06.004. PMID 20620037

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tiotropium | Placebo
Started | 1989 | 2002
Completed | 1671 | 1629
Not Completed | 318 | 373
Not completed — Adverse Event | 143 | 156
Not completed — Protocol Violation | 47 | 35
Not completed — Withdrawal by Subject | 20 | 35
Not completed — Lack of Efficacy | 28 | 67
Not completed — Lost to Follow-up | 22 | 28
Not completed — Other | 58 | 52

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium | Placebo | Total
Number analyzed (Participants) | 1952 | 1965 | 3917
Age, Continuous [Mean (Standard Deviation); unit: Years] — The TS was made up of all randomised and treated participants excluding 74 patients with potential fraudulent data from one investigator site
  Years | 64.8 (9.1) | 64.8 (9) | 64.80 (9.00)
Sex: Female, Male [Count of Participants; unit: Participants] — The TS was made up of all randomised and treated participants excluding 74 patients with potential fraudulent data from one investigator site
  Participants
    Female | 428 | 452 | 880
    Male | 1524 | 1513 | 3037

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) at Day 337
Description: Trough FEV1 is defined as the FEV1 measured at the -10 min time point at the end of the dosing interval (24 h post drug administration).
Time Frame: Baseline and Day 337
Population: The FAS was made up of all randomised and treated participants excluding 99 patients with questionable data. 133 participants from the FAS were excluded due to insufficient FEV1 data.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1889 | 1870
Litres | 0.119 (0.007) | 0.018 (0.007)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA with pooled centre, LABA use, and treatment fitted as main effects and the baseline trough FEV1 as a covariate; Mean Difference (Final Values) = 0.102, 95% CI 2-sided [0.085 to 0.118], Standard Error of Mean 0.009

2. Primary Outcome: Time to First Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: Time to first COPD exacerbation (defined as a complex of respiratory events/symptoms (increase or new onset) with a duration of 3 days or more requiring a change in treatment). Time is days from start of study treatment to onset of exacerbation.
Time Frame: During actual study treatment period (planned Day 1 to Day 337)
Population: The FAS was made up of all randomised and treated participants excluding 99 patients with questionable data.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1939 | 1953
Days | NA [NA to NA] — As <50% of the patients experienced an exacerbation in both treatment groups the median and 95% confidence interval were not estimable. Refer to the secondary endpoint 'Number of patients with at least one COPD exacerbation' for further information. | NA [354.0 to NA] — As <50% of the patients experienced an exacerbation in both treatment groups the median and 95% confidence interval were not estimable. Refer to the secondary endpoint 'Number of patients with at least one COPD exacerbation' for further information.

3. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) at Day 29
Description: Trough FEV1 is the mean volume of air that can be forced out in one second after taking a deep breath approximately 24 hours after the last administration of study drug.
Time Frame: Baseline and Day 29
Population: The FAS was made up of all randomised and treated participants excluding 99 patients with questionable data. 147 participants from the FAS were excluded due to insufficient FEV1 data.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1879 | 1866
Litres | 0.11 (0.005) | 0.017 (0.005)

4. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) at Day 169
Description: as for outcome 3
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1889 | 1870
Litres | 0.121 (0.006) | 0.018 (0.006)

5. Secondary Outcome: Number of COPD Exacerbations Per Patient - Exposure Adjusted
Description: Number of COPD exacerbations (defined as a complex of respiratory events/symptoms (increase or new onset) with a duration of 3 days or more requiring a change in treatment) per patient adjusted by length of treatment exposure (i.e. number of exacerbations multiplied by 365.25 and then divided by days of treatment exposure)
Time Frame: During actual study treatment period (planned Day 1 to Day 337)
Population: The FAS was made up of all randomised and treated participants excluding 99 patients with questionable data.
Measure: Median (Full Range); unit: COPD exacerbations per year
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1939 | 1953
COPD exacerbations per year | 0 (0) [0 to 21.5] | 0 (0) [0 to 182.6]

6. Secondary Outcome: Number of COPD Exacerbations Per Patient - naïve Estimate
Description: Number of COPD exacerbations (defined as a complex of respiratory events/symptoms (increase or new onset) with a duration of 3 days or more requiring a change in treatment) per patient not adjusted for treatment exposure (i.e. naïve estimate)
Time Frame: During actual study treatment period (planned Day 1 to Day 337)
Population: The FAS was made up of all randomised and treated participants excluding 99 patients with questionable data.
Measure: Median (Full Range); unit: COPD exacerbations
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1939 | 1953
COPD exacerbations | 0 (0) [0 to 9] | 0 (0) [0 to 10]

7. Secondary Outcome: Number of Patients With at Least One COPD Exacerbation
Description: Number of patients with at least one COPD exacerbation (defined as a complex of respiratory events/symptoms (increase or new onset) with a duration of 3 days or more requiring a change in treatment)
Time Frame: During actual study treatment period (planned Day 1 to Day 337)
Population: The FAS was made up of all randomised and treated participants excluding 99 patients with questionable data.
Measure: Number; unit: participants
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1939 | 1953
participants | 685 | 842

8. Secondary Outcome: Time to First Hospitalisation for COPD Exacerbation
Description: Time to first hospitalisation for COPD exacerbation (a complex of respiratory events/symptoms (increase or new onset) with a duration of 3 days or more requiring a change in treatment). Time is days from start of study treatment to onset of exacerbation
Time Frame: During actual study treatment period (planned Day 1 to Day 337)
Population: The FAS was made up of all randomised and treated participants excluding 99 patients with questionable data.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1939 | 1953
Days | NA [NA to NA] — As <50% of the patients experienced an exacerbation in both treatment groups the median and 95% confidence interval were not estimable. Refer to the secondary endpoint 'Number of patients with at least one COPD exacerbation' for further information. | NA [NA to NA] — As <50% of the patients experienced an exacerbation in both treatment groups the median and 95% confidence interval were not estimable. Refer to the secondary endpoint 'Number of patients with at least one COPD exacerbation' for further information.

9. Secondary Outcome: Number of Hospitalisations for COPD Exacerbations Per Patient - Exposure Adjusted
Description: Number of hospitalisations for COPD exacerbations (a complex of respiratory events/symptoms (increase or new onset) with a duration of 3 days or more requiring a change in treatment) per patient adjusted by length of treatment exposure (i.e. no. of exacerbations multiplied by 365.25 and then divided by days of treatment exposure)
Time Frame: During actual study treatment period (planned Day 1 to Day 337)
Population: The FAS was made up of all randomised and treated participants excluding 99 patients with questionable data.
Measure: Median (Full Range); unit: hospitalisations for COPD exacerbations
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1939 | 1953
hospitalisations for COPD exacerbations | 0 (0) [0 to 21.5] | 0 (0) [0 to 91.3]

10. Secondary Outcome: Number of Hospitalisations for COPD Exacerbations Per Patient - naïve Estimate
Description: Number of hospitalisations for COPD exacerbations (a complex of respiratory events/symptoms (increase or new onset) with a duration of 3 days or more requiring a change in treatment) per patient not adjusted for treatment exposure (i.e. naïve estimate)
Time Frame: During actual study treatment period (planned Day 1 to Day 337)
Population: The FAS was made up of all randomised and treated participants excluding 99 patients with questionable data.
Measure: Median (Full Range); unit: hospitalisations for COPD exacerbations
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1939 | 1953
hospitalisations for COPD exacerbations | 0 (0) [0 to 5] | 0 (0) [0 to 4]

11. Secondary Outcome: Number of Patients With at Least One Hospitalisation for a COPD Exacerbation
Description: Number of patients with at least one hospitalisation for a COPD exacerbation (a complex of respiratory events/symptoms (increase or new onset) with a duration of 3 days or more requiring a change in treatment)
Time Frame: During actual study treatment period (planned Day 1 to Day 337)
Population: The FAS was made up of all randomised and treated participants excluding 99 patients with questionable data.
Measure: Number; unit: participants
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1939 | 1953
participants | 161 | 198

12. Secondary Outcome: Change From Baseline in Saint George's Respiratory Questionnaire (SGRQ) Total Score at Day 337
Description: The SGRQ total score measures quality of life on a continuous scale ranging from 0=best state to 100=worst state
Time Frame: Baseline and Day 337
Population: The FAS was made up of all randomised and treated participants excluding 99 patients with questionable data. 534 participants from the FAS were excluded due to insufficient SGRQ data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1690 | 1668
Units on a scale | -4.726 (0.372) | -1.787 (0.374)

13. Secondary Outcome: Change From Baseline in Saint George's Respiratory Questionnaire (SGRQ) Total Score at Day 169
Description: The SGRQ total score measures quality of life on a continuous scale ranging from 0=best state to 100=worst state
Time Frame: Baseline and Day 169
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1690 | 1668
Units on a scale | -4.764 (0.348) | -2.568 (0.35)

14. Secondary Outcome: Change From Baseline in Saint George's Respiratory Questionnaire (SGRQ) Domain Score at Day 337
Description: The SGRQ domain score (symptom, activity and impact) measures quality of life on a continuous scale ranging from 0=best state to 100=worst state
Time Frame: Baseline and Day 337
Population: The FAS was made up of all randomised and treated participants excluding 99 patients with questionable data. Up to 534 participants from the FAS were excluded due to insufficient SGRQ data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1939 | 1953
Units on a scale
  Symptoms (N=1704,1688) | -7.260 (0.546) | -3.307 (0.548)
  Activities (N=1690,1668) | -3.196 (0.456) | -0.226 (0.460)
  Impacts (N=1690,1668) | -4.873 (0.409) | -2.038 (0.412)

15. Secondary Outcome: Change From Baseline in Saint George's Respiratory Questionnaire (SGRQ) Domain Score at Day 169
Description: as for outcome 14
Time Frame: Baseline and Day 169
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1939 | 1953
Units on a scale
  Symptoms (N=1704,1688) | -6.555 (0.530) | -3.268 (0.532)
  Activities (N=1690,1668) | -3.573 (0.432) | -1.218 (0.435)
  Impacts (N=1690,1668) | -4.917 (0.390) | -2.935 (0.392)

16. Secondary Outcome: Change From Baseline in Trough Forced Vital Capacity (FVC) at Day 29
Description: Trough FVC is the mean maximum volume of air that can be forcibly expired from the lungs; measured approximately 24 hours after the last administration of study drug.
Time Frame: Baseline and Day 29
Population: The FAS was made up of all randomised and treated participants excluding 99 patients with questionable data. 147 participants from the FAS were excluded due to insufficient FVC data.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1879 | 1866
Litres | 0.176 (0.009) | 0.025 (0.009)

17. Secondary Outcome: Change From Baseline in Trough Forced Vital Capacity (FVC) at Day 169
Description: as for outcome 16
Time Frame: Baseline and Day 169
Population: The FAS was made up of all randomised and treated participants excluding 99 patients with questionable data. 133 participants from the FAS were excluded due to insufficient FVC data.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1889 | 1870
Litres | 0.179 (0.010) | 0.019 (0.010)

18. Secondary Outcome: Change From Baseline in Trough Forced Vital Capacity (FVC) at Day 337
Description: as for outcome 16
Time Frame: Baseline and Day 337
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1889 | 1870
Litres | 0.168 (0.011) | -0.001 (0.011)

19. Secondary Outcome: Marked Changes From Baseline in Vital Signs at End of Treatment
Description: Marked changes from baseline in vital signs (diastolic and systolic blood pressure (DBP and SBP) and pulse rate (PR)) at end of treatment.
  SBP - Increase means SBP >150 mmHg and an increase above baseline of >25 mmHg. SBP - Decrease means SBP <100 mmHg and a decrease below baseline of >10 mmHg.
  DBP - Increase means DBP >90 mmHg and an increase above baseline of >10 mmHg. DBP - Decrease means DBP <60 mmHg and a decrease below baseline of >10 mmHg.
  PR - Increase means PR >100 bpm and an increase above baseline of >10 bpm. PR - Decrease means PR <60 bpm and a decrease below baseline of >10 bpm.
Time Frame: Baseline and end of treatment
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1747 | 1749
participants
  SBP - Increase | 29 | 31
  SBP - Decrease | 6 | 12
  DBP - Increase | 40 | 39
  DBP - Decrease | 9 | 14
  PR - Increase | 35 | 43
  PR - Decrease | 26 | 26

20. Secondary Outcome: Clinically Relevant Findings in Physical Examination and ECG
Description: Clinically relevant findings in Physical Examination and ECG at end of treatment
Time Frame: End of treatment
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 1952 | 1965
participants
  Phys. Exam - No new/worsened finding | 1723 | 1733
  Phys. Exam - new or worsened finding | 22 | 17
  Phys. Exam - Missing | 207 | 215
  ECG - No new/worsened finding | 1674 | 1677
  ECG - new or worsened finding | 37 | 39
  ECG - Missing | 241 | 249

ADVERSE EVENTS:
Time Frame: From first drug administration until 30 days after last drug administration.
Description: 74 patients were excluded from the treated set due to potential fraudulent data from one investigator site
Arm/Group | Tiotropium | Placebo
Serious Adverse Events (participants affected / at risk) | 342/1952 | 336/1965
Other Adverse Events (participants affected / at risk) | 866/1952 | 926/1965
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium (N=1952) | Placebo (N=1965)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 3 | 2
Acute myocardial infarction (Cardiac disorders) | 2 | 5
Angina pectoris (Cardiac disorders) | 4 | 3
Angina unstable (Cardiac disorders) | 1 | 5
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 2 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 2
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 8 | 10
Cardiac failure congestive (Cardiac disorders) | 5 | 4
Cardiac valve disease (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 4 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Cor pulmonale (Cardiac disorders) | 2 | 3
Cor pulmonale acute (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 5 | 2
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 2 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 5 | 5
Myocardial ischaemia (Cardiac disorders) | 5 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 1
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Tricuspid valve disease (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Chilaiditi's syndrome (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 5
Duodenal ulcer (Gastrointestinal disorders) | 0 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 6 | 6
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 2 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Proctocolitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 2
Umbilical hernia (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Volvulus (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 1
Chest discomfort (General disorders) | 2 | 0
Chest pain (General disorders) | 4 | 0
Death (General disorders) | 5 | 1
Drowning (General disorders) | 2 | 0
Drug interaction (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Mass (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 2 | 1
Pitting oedema (General disorders) | 0 | 1
Polyp (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Sudden death (General disorders) | 2 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecysititis (Hepatobiliary disorders) | 1 | 1
Cholecysititis acute (Hepatobiliary disorders) | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Abscess intestinal (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 7 | 6
Bronchopneumonia (Infections and infestations) | 2 | 4
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Bursitis infective (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 1
Empyema (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Epiglottitis haemophilus (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 6
Gastroenteritis viral (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 3
Infection (Infections and infestations) | 0 | 2
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 9 | 18
Influenza (Infections and infestations) | 0 | 2
Lobar pneumonia (Infections and infestations) | 3 | 7
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 6
Lung infection (Infections and infestations) | 0 | 2
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 0 | 1
Pharyngeal abscess (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 26 | 37
Postoperative wound infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 4 | 2
Septic shock (Infections and infestations) | 2 | 2
Staphylococcal infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract infection fungal (Infections and infestations) | 1 | 0
Accident (Injury, poisoning and procedural complications) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 4
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 3 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 4 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alcohol increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 1
Blood pressure increased (Investigations) | 1 | 0
Chest x-ray abnormal (Investigations) | 1 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 0
Diabetic foot (Metabolism and nutrition disorders) | 2 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Benigh neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Hypopharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 2
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ataxia (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebral circulatory failure (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 3 | 2
Cerebral thrombosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Cervical myelopathy (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2
Dysarthria (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 1
Lethargy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 1
Monoparesis (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Syncope vasovagal (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 3
Unresponsive to stimuli (Nervous system disorders) | 1 | 0
Vascular dementia (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 2
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 2 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 1
Renal failure acute (Renal and urinary disorders) | 3 | 2
Urethral meatus stenosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 5 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 6 | 3
Prostatic haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 130 | 155
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lichen nitidus (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Living in residential institution (Social circumstances) | 1 | 0
Gallbladder operation (Surgical and medical procedures) | 1 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 1
Ileostomy closure (Surgical and medical procedures) | 1 | 0
Shoulder arthroplasty (Surgical and medical procedures) | 0 | 1
Urethrotomy (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 2 | 2
Aortic rupture (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Arterial stenosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 2
Hypovolaemic shock (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Venous insufficiency (Vascular disorders) | 0 | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium (N=1952) | Placebo (N=1965)
Nasopharyngitis (Infections and infestations) | 157 | 151
Upper respiratory tract infection (Infections and infestations) | 97 | 123
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 561 | 659
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 122 | 144
Cough (Respiratory, thoracic and mediastinal disorders) | 123 | 106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.